CLINICAL TRIAL: NCT07228026
Title: A Combined Prospective, Multicenter, Non-Randomized, Open-Label, Point-of-Care and Home Use Pivotal Study of the fenoTRACK Device for Monitoring Changes of Fractional Exhaled Nitric Oxide (FeNO) in Non-Steroid-Treated Adult and Pediatric Uncontrolled Asthma Subjects and a Prospective Multicenter Clinical Precision Evaluation for Point-of-Care and Home Use in Adult and Pediatric Controlled Asthma Subjects
Brief Title: Use of fenoTRACK Device for Monitoring Changes of Fractional Exhaled Nitric Oxide (FeNO) in Uncontrolled Asthma Subjects and Controlled Asthma Subjects
Status: Recruiting | Type: Observational
Sponsor: Biometry Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: F1
Record Dates: First submitted 2025-10-27; First posted 2025-11-13 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: Asthma; FeNO
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uncontrolled Asthma Subjects: fenoTRACK for Uncontrolled Adult and Pediatric Asthma Subjects
  Interventions: Device: fenoTRACK Device
- Controlled Asthma Subjects: fenoTRACK for Controlled Adult and Pediatric Asthma Subjects
  Interventions: Device: fenoTRACK Device

INTERVENTIONS:
Device: fenoTRACK Device — Home FeNO Monitoring: FeNO measurement will be performed.
  POC Longitudinal Response to Treatment: FeNO measurement will be performed in the office both the simulated home environment and POC environment.

SUMMARY:
This study incorporates objectives directed at two subject cohorts:

1. Uncontrolled Adult and Pediatric Asthma Subjects: To demonstrate a statistically significant and clinically meaningful decline in Point Of Care (POC) FeNO as measured by the fenoTRACK device, after an approximately 2-week course of corticosteroid therapy in adults and children with non-steroid treated uncontrolled asthma.
2. Controlled Adult and Pediatric Asthma Subjects:

   * To evaluate within-session clinical precision during Visit 1 and Visit 2 for the fenoTRACK device for simulated at home FeNO, and at POC
   * To evaluate within-session clinical precision for home fenoTRACK use

DETAILED DESCRIPTION:
1. Uncontrolled Adult and Pediatric Asthma Subjects The primary objective is: To demonstrate a statistically significant and clinically meaningful decline in POC FeNO as measured by the fenoTRACK device from Visit 1 (V1) to Visit 2 (V2), after an approximately 2-week course of corticosteroid therapy in adults and children with non-steroid treated uncontrolled asthma.

   Secondary objectives:
   * To demonstrate that the decline in FeNO on the fenoTRACK device is accompanied by improvements in asthma outcome measures including the 7-item asthma control questionnaire (ACQ) score or asthma control questionnaire - Interviewer Administered (ACQ-IA), lung function as assessed by spirometry, and rescue medication use
   * To demonstrate clinical accuracy of FeNO measurements on the fenoTRACK device by comparison of within-session FeNO values acquired in a simulated at home FeNO versus FeNO values acquired at the POC at V1 and V2
   * To record how many efforts are required to achieve 2 valid FeNO results on the fenoTRACK device for simulated at home FeNO and POC FeNO measurements at V1 and V2, and between V1 and V2
2. Controlled Adult and Pediatric Asthma Subjects

Co-primary objectives:

* To evaluate within-session clinical precision during V1 and V2 for the fenoTRACK device for simulated at home FeNO, and at POC To evaluate within-session clinical precision for home fenoTRACK use Secondary objectives:To demonstrate clinical accuracy of FeNO measurements on the fenoTRACK device by comparison of within-session FeNO values acquired for simulated at home FeNO versus FeNO values acquired at the POC at V1 and V2
* To record how many efforts are required to achieve 2 valid FeNO results on the fenoTRACK device for simulated at home FeNO and POC measurements at V1 and V2, and between V1 and V2

ELIGIBILITY:
Inclusion Criteria Uncontrolled Cohort:

1. The subject is male or female age 5 years and above
2. The subject and/or their Legally Authorized Representative (LAR) in the case of a minor has signed an Informed Consent Form (ICF) and Assent (as applicable per IRB requirements) and understands the risks and benefits of the study
3. The subject has a diagnosis of asthma
4. The subject is willing and able to perform all study procedures
5. The subject must have uncontrolled asthma as defined by the presence on at least 2 days per week (can be non-consecutive days) in the 7 days prior to V1 of at least 3 symptoms from the following list:

   i. Cough ii. Wheezing iii. Shortness of breath iv. Chest tightness v. Nocturnal awakening with asthma vi. Limitation in activity due to asthma
6. The subject has a FeNO value based on the first measurement of at least 30 ppb if an adult or at least 25 ppb if <18 years old measured on a cleared FeNO device (e.g., NIOX VERO®)

Inclusion Criteria Controlled Cohort:

1. The subject is male or female age 5 years and above
2. The subject and/or their Legally Authorized Representative (LAR) in the case of a minor has signed an Informed Consent Form (ICF) and Assent (as applicable per IRB requirements) and understands the risks and benefits of the study
3. The subject has an established diagnosis of asthma for at least 180 days prior to V1
4. The subject is willing and able to perform all study procedures

Exclusion Criteria Uncontrolled:

1. The subject is in need of immediate referral to the emergency department
2. The subject has taken the following medications in the indicated period before V1:

   1. OCS within 4 weeks
   2. ICS within 2 weeks
   3. Biologic therapies (e.g., omalizumab or dupilumab) within 12 weeks. Note: Use of as needed ICS+SABA is also exclusionary in the 2 weeks prior to V1
3. The subject has a contraindication to corticosteroids.
4. The subject has demonstrated significant non-compliance during a previous clinical trial
5. The subject participated in any clinical study involving a drug, biologic, or device within 30 days prior to V1 or within 5 half-lives for drugs, whichever duration is shorter
6. The subject has other significant respiratory conditions, e.g., Chronic Obstructive Pulmonary Disease, cystic fibrosis
7. Subject is an employee/relative of the following:

   1. Biometry Inc.
   2. Contract Research Organization(s) running the study
   3. Investigational Site
   4. Study Vendors
8. Any other condition(s), that in the Investigator's opinion, make it undesirable for the subject to participate in the study
9. A ≥ 10 pack-year history of smoking or smoking in the 180 days prior to V1 (pack years = average packs/day x years of exposure) Note: smoking includes cigarettes, electronic cigarettes, cigars, and chewing or dipping tobacco
10. Pregnant or nursing subjects

Exclusion Criteria Controlled:

1. The subject has other significant respiratory conditions, e.g., Chronic Obstructive Pulmonary Disease, cystic fibrosis
2. The subject has demonstrated significant non-compliance during a previous clinical trial
3. The subject participated in any clinical study involving a drug, biologic, or device within 30 days prior to V1 or within 5 half-lives for drugs, whichever duration is shorter.
4. Subject is an employee/relative of the following:

   1. Biometry Inc.
   2. Contract Research Organization(s) running the study
   3. Investigational Site
   4. Study Vendors
5. Any other condition(s), that in the Investigator's opinion, make it undesirable for the subject to participate in the study
6. A ≥ 10 pack-year history of smoking or smoking in the 180 days prior to V1 (pack years = average packs/day x years of exposure) Note: smoking includes cigarettes, electronic cigarettes, cigars, and chewing or dipping tobacco
7. Pregnant or nursing subjects

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes two distinct cohorts. The first cohort comprises male and female subjects aged 5 and above with uncontrolled asthma (See uncontrolled Asthma subject Inclusion Criteria). The second cohort comprises male and female subjects aged 5 and above with controlled asthma. If one of the subject cohorts completes before the other, the Sponsor reserves the right to analyze that cohort first.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Uncontrolled Cohort - Magnitude of change in FeNO Values | Visit 2 (Day 14)
  Magnitude of change, expressed both as absolute and percentage change in FeNO values in the uncontrolled cohort from Visit 1 to Visit 2.

SECONDARY OUTCOMES:
Uncontrolled Cohort - Magnitude of change (POC) | Visit 2 (Day 14)
  Magnitude of change expressed both as absolute and percentage change, in POC FeNO values using the fenoTRACK device in the uncontrolled cohort.
Uncontrolled Cohort - Magnitude of change (Home Use) | Day 1 and Day 2 AM and PM FeNO values compared to average of the last 2 Days prior to Visit 2
  Uncontrolled Cohort - Magnitude of change expressed both as absolute and percentage change, in actual at home using the fenoTRACK device in the uncontrolled cohort.
Uncontrolled Cohort - Change in 7-item ACQ/ACQ-IA | Visit 2 (Day 14)
  The changes in 7-item ACQ/ACQ-IA Scores for both questionnaires from V1 to V2 will be estimated in the uncontrolled Cohort
Uncontrolled Cohort - Change in best spirometry measures | Visit 2 (Day 14)
  Change in best spirometry measures, both absolute and percent, Forced Expiratory Volume (FEV1), Forced Vital Capacity (FVC), FEV1/FVC in the uncontrolled cohort.
Controlled cohort - Clinical precision based on the first 2 FeNO results - Within-session clinical precision in a simulated home-use environment (V1 and V2) - Within-session clinical precision at the POC (V1 and V2) - Clinical precision at home | Visit 2 (Day 14)
  Precision is assessed by evaluating the statistical repeatability of two exhaled nitric oxide (FeNO) measurements which are measured by the fenoTRACK investigational device in parts per billion. This will be assessed at Visit 1 and Visit 2 using the Simulated at home, POC and at home setting in the controlled cohort.
Controlled cohort - Accuracy of FeNO results by comparison of paired within-individual FeNO values acquired in a simulated home-use environment versus FeNO values acquired at the POC at both V1 and V2 | Visit 2 (Day 14)
  Accuracy for a diagnostic measure means that the FeNO values in parts per billion measured by the fenoTRACK investigational device will be compared statistically between the simulated at home i.e. independently acquired measures and the POC measures obtained under supervision in the clinic. Accuracy is expressed as a correlation value and confidence limits for the correlation between the two measures in the controlled cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Philip E. Silkoff, MD, Principal Investigator — Precision ClinOps LLC
Locations (13):
- United States (13):
  - Bensch Clinical Research LLC, Stockton, California
  - AllerVie Clinical Research, Panama City, Florida
  - AllerVie Clinical Research, Columbus, Georgia
  - Paul A Shapero MD, Bangor, Maine
  - AllerVie Clinical Research, Ellicott City, Maryland
  - AllerVie Clinical Research, Glenn Dale, Maryland
  - Nebraska Medical Research Institute, Inc., Bellevue, Nebraska
  - Allergy Partners Clinical Research, Asheville, North Carolina
  - Toledo Institute of Clinical Research Inc, Toledo, Ohio
  - Orion Clinical Research, Austin, Texas
  - Pharmaceutical Research & Consulting, Inc., Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Allergy, Asthma & Sinus Center, S.C., Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No